CLINICAL TRIAL: NCT05167799
Title: Cardiac Contractility Modulation Therapy in Amyloid Cardiomyopathy Patients With Heart Failure With Mid-range Ejection Fraction: a Multicentre Registry
Brief Title: Cardiac Contractility Modulation Therapy in Amyloid Cardiomyopathy Patients With Heart Failure
Acronym: AMY-CCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale C & G Mazzoni (Other)
Responsible Party: Principal Investigator, Procolo Marchese, Principal Investigator, Ospedale C & G Mazzoni
Other Study IDs: AMYCCM190421
Record Dates: First submitted 2021-12-07; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Amyloidosis Cardiac; Heart Failure
Keywords: Cardiac Amyloidosis; Heart Failure; Cardiac Contractility Modulation; CCM
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Amyloidosis patients: Patients with established diagnosis of amyloid TTR Cardiomyopathy, baseline ejection fraction ≥25% and ≤45%, at least one hospitalization due to worsening heart failure over the year before entry into the registry.
  Already implanted with ICD or PM if needed, fullfilling the indication for CCM implantation.
  Interventions: Device: Cardiac Contractility Modulation (CCM)

INTERVENTIONS:
Device: Cardiac Contractility Modulation (CCM) — Patients will be implanted with CCM device according to indications, to improve Heart Failure symptoms and then enrolled in the Registry if they fullfil Inclusion and Exclusion Criteria (First of all if they are diagnosed with TTR Amyloidosis)

SUMMARY:
The primary aim of this observational registry is to evaluate the efficacy of CCM in patients with heart failure with mid-range or reduced EF and diagnosis of TTR amyloidosis. The efficacy will be evaluated in terms of composite of occurrence of heart failure-related hospitalizations and/or acute intravenous interventions (IVI) at 12-month follow up compared to those reported 12 months before CCM implantation. Among the secondary endpoints, clinical functional status, quality of life, drug changes and Echocardiographic parameters will be evaluated and compared from baseline to follow up.

DETAILED DESCRIPTION:
Amyloidosis represents a group of human degenerative diseases characterized by the deposition of aggregates of abnormally folded proteins in single or multi-organs. Cardiac amyloidosis is primarily associated with the systemic production and release of a number of amyloidogenic proteins, notably immunoglobulin light chain proteins (also known as amyloid light chain or AL) or transthyretin proteins (TTR). Notably, although myocardial dysfunction is generally understood as a result of infiltration by extracellular amyloid deposits, there is experimental evidence of direct cytotoxic effect, possibly due to oxidative stress.

Since neither HF optimal medical therapy nor HF devices seems to have a clear benefit in amyloid cardiomyopathy, this clinical setting needs to test other therapeutic options.

Randomized clinical trials have shown that Cardiac contractility modulation (CCM) may be considered as a concrete therapeutic option in patients with symptomatic Heart Failure (HF) despite optimal medical therapy (OMT), with Left Ventricular Ejection Fraction (LVEF) between 25% and 45%, with narrow QRS complex (<130ms).

CCM signal treatment reverses the cardiac maladaptive fetal gene program and normalizes expression of key sarcoplasmic reticulum Ca2+ cycling and stretch response genes. Specifically, 3-month on CCM therapy resulted in decreased expression of A- and B-type natriuretic peptides, p38 mitogen activated protein kinase (MAPK) and p21 Ras and increased expression of α-MHC, SERCA-2a, phospholamban, and ryanodine receptors. Notably, pre-clinical data suggest that triggering p38α MAPK autophosphorylation plays a crucial role in amyloidogenic light-chain mediated cellular oxidative stress, dysfunction and ultimately cell death in cardiomyocytes. Therefore CCM mechanism of action could be beneficial in cardiac amyloidosis but there are no data in this specific clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Male or a nonpregnant female
* All of the following: Established diagnosis of amyloid TTR Cardiomyopathy; baseline ejection fraction ≥25% and ≤45%; at least one hospitalization due to worsening heart failure over the year before entry into the registry.
* ICD if indicated
* PM if indicated
* Willing and able to return for all follow-up visits

Exclusion Criteria:

* AL amyloid cardiomyopathy
* Subjects who have a potentially correctible cause of heart failure (eg, Ischemic or valvular or congenital heart disease).
* Scheduled for CABG or PCI or has undergone a CABG within 90 d or PCI within 30 d.
* Myocardial infarction within 90 days
* Mechanical tricuspid valve
* Prior heart transplant
* Chronic haemodialysis
* Familial TTR amyloidotic cardiomyopathy with significant polyneuropathy potentially eligible for Patirisan or Inotersen17
* Unable to provide informed consent

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This Registry includes patients with chronic, symptomatic heart failure with moderately-to-severely reduced left ventricular systolic function despite optimal pharmacological and electrical therapy, who have been diagnosed with TTR Cardiac Amyloidosis. The clinical trial study (prospective registry) will be conducted in accordance with the protocol, with the Helsinki Declaration and with the favorable opinion of the local Ethics Committee of the participating Centers.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite of occurrence of hospitalizations due to worsening of heart failure and/or acute intravenous administrations of diuretics or inotropic drugs over the 12 months after entry into the registry. | 12-month
  The occurrence of any of the events mentioned (worsening of heart failure or intravenous intervention) involves reaching the endpoint

SECONDARY OUTCOMES:
Occurrence of clinical need to increase oral dose of diuretic drug and/or to add another diuretic drug class | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month
Occurrence of oral dose diuretic drug reduction | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month
NYHA class | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month
Distance walked at the 6-minute walking test | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month in meters walked during the test
Kansas City Cardiomyopathy Questionnaire-Overall Summary (KCCQ-OS) score | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month in the KCCQ-OS score
Biomarker (NT-proBNP) | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month in the biomarker level (pg/ml)
Biomarker (HS-Troponin) | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month in the biomarker level (ng/l)
Echocardiographic parameters (Ejection Fraction) | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month in EF (%)
Echocardiographic parameters (End diastolic volume and End systolic volume) | 12-month
  Change from baseline to 2 weeks, 1,3, 6 and 12-month in End diastolic volume and End systolic volume respectively (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Procolo Marchese, MD, Principal Investigator — Ospedale Mazzoni (Ascoli Piceno)
Locations (1):
- Ospedale Mazzoni, Ascoli Piceno, Marche (AP), Italy

REFERENCES:
- [Result] Shi J, Guan J, Jiang B, Brenner DA, Del Monte F, Ward JE, Connors LH, Sawyer DB, Semigran MJ, Macgillivray TE, Seldin DC, Falk R, Liao R. Amyloidogenic light chains induce cardiomyocyte contractile dysfunction and apoptosis via a non-canonical p38alpha MAPK pathway. Proc Natl Acad Sci U S A. 2010 Mar 2;107(9):4188-93. doi: 10.1073/pnas.0912263107. Epub 2010 Feb 11. PMID 20150510
- [Result] Brenner DA, Jain M, Pimentel DR, Wang B, Connors LH, Skinner M, Apstein CS, Liao R. Human amyloidogenic light chains directly impair cardiomyocyte function through an increase in cellular oxidant stress. Circ Res. 2004 Apr 30;94(8):1008-10. doi: 10.1161/01.RES.0000126569.75419.74. Epub 2004 Mar 25. PMID 15044325
- [Result] Kristen AV, Dengler TJ, Hegenbart U, Schonland SO, Goldschmidt H, Sack FU, Voss F, Becker R, Katus HA, Bauer A. Prophylactic implantation of cardioverter-defibrillator in patients with severe cardiac amyloidosis and high risk for sudden cardiac death. Heart Rhythm. 2008 Feb;5(2):235-40. doi: 10.1016/j.hrthm.2007.10.016. Epub 2007 Oct 9. PMID 18242546
- [Result] Abraham WT, Kuck KH, Goldsmith RL, Lindenfeld J, Reddy VY, Carson PE, Mann DL, Saville B, Parise H, Chan R, Wiegn P, Hastings JL, Kaplan AJ, Edelmann F, Luthje L, Kahwash R, Tomassoni GF, Gutterman DD, Stagg A, Burkhoff D, Hasenfuss G. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Cardiac Contractility Modulation. JACC Heart Fail. 2018 Oct;6(10):874-883. doi: 10.1016/j.jchf.2018.04.010. Epub 2018 May 10. PMID 29754812
- [Result] Anker SD, Borggrefe M, Neuser H, Ohlow MA, Roger S, Goette A, Remppis BA, Kuck KH, Najarian KB, Gutterman DD, Rousso B, Burkhoff D, Hasenfuss G. Cardiac contractility modulation improves long-term survival and hospitalizations in heart failure with reduced ejection fraction. Eur J Heart Fail. 2019 Sep;21(9):1103-1113. doi: 10.1002/ejhf.1374. Epub 2019 Jan 16. PMID 30652394